CLINICAL TRIAL: NCT07402278
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effects of Oral Intake of HB05P on Improving Muscle Strength
Brief Title: Evaluation of HB05P for Muscle Strength Improvement in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthbiome Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2404-009-597
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Age-Related Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB05P (Experimental): Pasteurized Akkermansia muciniphila HB05P, 3×10¹⁰ cells/day, once daily for 12 weeks
  Interventions: Dietary Supplement: HB05P (Pasteurized Akkermansia muciniphila)
- Placebo (Placebo Comparator): Placebo capsule containing crystalline cellulose, once daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HB05P (Pasteurized Akkermansia muciniphila) — Pasteurized Akkermansia muciniphila HB05P capsule containing 150mg HB05P (3×10¹⁰ cells/day). One capsule taken orally once daily after breakfast for 12 weeks (84 days).
  Arms: HB05P
Dietary Supplement: Placebo — Matching placebo capsule containing crystalline cellulose. One capsule taken orally once daily after breakfast for 12 weeks (84 days).
  Arms: Placebo

SUMMARY:
This study aims to clinically and scientifically evaluate the safety of HB05P intake as a functional ingredient for health functional foods, as well as its efficacy in improving muscle strength.

This study is designed as a randomized, double-blind, placebo-controlled trial. Subjects who voluntarily agree to participate in the study by providing written informed consent will be screened according to the inclusion and exclusion criteria. Subjects who are taking health functional foods or medications that are judged not to affect the study outcomes may continue their use during the study. Eligible subjects will be randomly assigned in a 1:1 ratio to either the test group or the control group.

Randomized subjects will be instructed to perform walking and resistance (muscle-strengthening) exercises at least three times per week, for 30 minutes to 1 hour per session, until the end of the study period. Subjects will be required to complete an exercise diary. They will also receive the investigational product and a daily intake diary, and will consume the study product once daily according to the instructed method.

The quality of life questionnaire (EQ-5D-5L), exercise diary, and dietary intake assessed using the 24-hour recall method will be evaluated and compared between baseline and post-intervention. Efficacy and safety assessment variables will be measured and tested at Day 0 and Day 84, and the collected data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or older and younger than 80 years (male or female) who meet the inclusion criteria and do not meet any exclusion criteria
* Body Mass Index (BMI) between 18.5 and 30.0 kg/m²
* Skeletal muscle mass less than 110% of standard value measured by Bioelectrical Impedance Analysis (BIA)
* Reduced handgrip strength in the dominant hand based on age- and sex-specific criteria: (Ages 60-69) Males ≤38.5 kg, Females ≤24.1 kg; (Ages 70-79) Males ≤33.2 kg, Females ≤20.9 kg
* Capable of normal physical activity and voluntarily providing written informed consent to participate in this study

Exclusion Criteria:

* History of bone fracture within the past 1 year
* Serum creatinine greater than 2 times the upper limit of normal at the study site
* AST (GOT) or ALT (GPT) greater than 2 times the upper limit of normal at the study site
* Current diabetes mellitus or fasting blood glucose ≥126 mg/dL
* Uncontrolled hyperthyroidism or hypothyroidism
* Uncontrolled hypertension (blood pressure ≥160/100 mmHg)
* Currently taking medication for psychiatric disorders (except for intermittent use for sleep disorders)
* Participation in another drug clinical trial within 1 month prior to screening
* Regular consumption (≥4 times/week) of probiotics or fermented dairy products (yogurt, cheese, etc.) within 2 weeks prior to screening
* Use of medications or health functional foods related to muscle function within 1 month prior to screening (refer to prohibited concomitant medications)
* History of gastrointestinal resection surgery (except appendectomy)
* Pregnant or lactating women, or women planning to become pregnant during the study period
* Known allergy to any component of the study product
* History of alcohol abuse
* Asthma or obstructive/restrictive pulmonary disease that may affect lung volume
* Uncooperative attitude or any condition that, in the investigator's judgment, would make the participant unsuitable for the study

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Isokinetic Knee Extension and Flexion Strength | Baseline and Week 12
  Change from baseline in isokinetic muscle strength of quadriceps and hamstrings (both left and right) measured by Biodex dynamometer at angular velocity of 60°/s

SECONDARY OUTCOMES:
Change in Isokinetic Muscle Power | Baseline and Week 12
  Change from baseline in muscle power measured by Biodex dynamometer at angular velocity of 60°/s
Change in Appendicular Skeletal Muscle Mass (ASM) | Baseline and Week 12
  Change from baseline in appendicular skeletal muscle mass measured by dual-energy X-ray absorptiometry (DEXA)
Change in Skeletal Muscle Mass Index (SMMI) | Baseline and Week 12
  Change from baseline in skeletal muscle mass index (ASM/height²) measured by DEXA
Change in Body Fat Percentage | Baseline and Week 12
  Change from baseline in total and trunk body fat percentage measured by DEXA
Change in Lower Extremity Muscle Mass | Baseline and Week 12
  Change from baseline in lower extremity muscle mass measured by DEXA
Change in Handgrip Strength | Baseline and Week 12
  Change from baseline in handgrip strength measured by hand dynamometer
Change in Short Physical Performance Battery (SPPB) Score | Baseline and Week 12
  Change from baseline in Short Physical Performance Battery (SPPB) total score (range 0-12; higher scores indicate better physical performance) and subscores: balance (0-4), gait speed (0-4), and chair stand (0-4)
Change in Serum IGF-1 Level | Baseline and Week 12
  Change from baseline in serum insulin-like growth factor-1 (IGF-1) concentration
Change in Serum Myostatin Level | Baseline and Week 12
  Change from baseline in serum myostatin concentration
Change in Serum Follistatin Level | Baseline and Week 12
  Change from baseline in serum follistatin concentration
Change in Serum Nutritional Markers | Baseline and Week 12
  Change from baseline in serum albumin, prealbumin, and total protein concentrations
Change in Health-Related Quality of Life | Baseline and Week 12
  Change from baseline in European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) index score (range -0.5 to 1.0; higher scores indicate better health-related quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Hyunlee Shin, MD, Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea